CLINICAL TRIAL: NCT04875234
Title: Vision Improvement for Legally Blind Dry Age-Related Macular Degeneration Patients
Brief Title: Vision Improvement for Legally Blind Dry AMD Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Optimal Acuity Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Retro3
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-04

CONDITIONS: Dry Age-related Macular Degeneration; Vision Impairment and Blindness
Keywords: AMD, vision impairment, blindness
MeSH Terms: conditions — Vision Disorders; Blindness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Legally Blind Dry AMD Patients: Legally Blind Dry AMD Patients with either unilateral or bilateral blindness
  Interventions: Device: Clear-K Low Vision Aid Treatment

INTERVENTIONS:
Device: Clear-K Low Vision Aid Treatment — A Clear-K Low Vision Aid Device is used to produce small corneal shape and refraction changes in order to redirect light onto functional areas of the retina.

SUMMARY:
This retrospective observational study is intended to assess the feasibility of using a nonsignificant risk device for vision improvement for legally blind dry AMD patients.

DETAILED DESCRIPTION:
This retrospective observational study is intended to assess the feasibility of using a nonsignificant risk device for vision improvement for legally blind dry Age-Related Macular Degneration patients. 12-month follow-up examinations will be used to assess the amount of vision improvement and its dependence on device parameters.

ELIGIBILITY:
IInclusion Criteria:

* Male or Female
* Any race
* Patient is at least 50 years old.
* Patient must have dry AMD in the study eye.
* Patient is legally blind due to AMD - i.e., has corrected distance visual acuity (CDVA) of 20/125 or worse (45 letters; logMAR ≥ 0.80) in the study eye.
* Patient has normal corneal surface topography on videokeratography (i.e., without distorted or unclear corneal mires).
* Patient is not a contact lens wearer.
* Patient is willing and able to comply with all examinations.
* Patient must be competent to sign an informed consent form before study entry.

Exclusion Criteria:

* Visually significant cataract in the study eye
* Presence of a visually significant posterior capsule opacity if prior cataract surgery has been performed in the study eye
* Any visually significant disease process in any ocular structure other than AMD that would affect vision in the study eye
* Previous corneal surgery in the study eye
* Presence or history of any other condition or finding that, in the opinion of the investigator, makes the patient unsuitable as a candidate for study participation or may confound the outcome of the study

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with dry age-related macular degeneration an legal blindness in one or both eyes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Best spectacle-corrected distance visual acuity (BCDVA) | 12 months post-treatment
  BCDVA measured using ETDRS eye charts

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berry, PhD, Principal Investigator — Optimal Acuity Corporation

IPD SHARING:
Plan to Share IPD: Undecided
Undecided